CLINICAL TRIAL: NCT02364362
Title: Docetaxel Plus Famitinib Versus Docetaxel Plus Placebo in Patients With Advanced Non-squamous and Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Study of Famitinib Plus Docetaxel in Patients With Advanced Non-squamous and Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-FMTN- Ⅱ-NSCLC-COM
Record Dates: First submitted 2015-01-19; First posted 2015-02-18 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2018-12

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Famitinib + docetaxel (Experimental): Low, medium and high dose of famitinib and 60 mg/m^2 docetaxel every 3 weeks
  Interventions: Drug: famitinib L + docetaxel; Drug: famitinib M + docetaxel; Drug: famitinib H + docetaxel

INTERVENTIONS:
Drug: famitinib L + docetaxel — famitinib 15mg qd + docetaxel 60 mg/m^2
Drug: famitinib M + docetaxel — famitinib 20mg qd + docetaxel 60 mg/m^2
Drug: famitinib H + docetaxel — famitinib 25mg qd + docetaxel 60 mg/m^2

SUMMARY:
Famitinib is a tyrosin-inhibitor agent targeting at c-Kit, VEGFR2, PDGFR, VEGFR3, Flt1 and Flt3. Phase I study has shown that the toxicity is manageable.

This study assessed the safety and maximum tolerated dose of continuous daily treatment with Famitinib plus docetaxel (60 mg/m^2, every 3 weeks) in patients with Advanced Non-squamous and Non-Small Cell Lung Cancer (NSCLC) to determine the recommended dose for the Phase II trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-70 years;
2. ECOG PS (Eastern Cooperative Oncology Group Performance Status)of 0 or 1;
3. Life expectancy of at least 12 weeks;
4. Histologically or cytologically confirmed, locally advanced and/or metastatic NSCLC of stage IIIB or IV or recurrent NSCLC;
5. Relapse or failure of one first line prior platinum-based chemotherapy;EGFR mutation type previously treated with platinum-based chemotherapy and EGFR inhibitors;
6. At least one target tumour lesion that has not been irradiated within the past 3 months and that can accurately be measured ,according to RECIST 1.1;
7. Participants have adequate organ and marrow function as defined below:

   * Hemoglobin ≥ 90g/L ( no blood transfusion in 2 weeks)
   * Absolute neutrophil count (ANC) ≥ 1.5×10^9/L
   * Platelets(PLT)≥ 100×10^9/L
   * Bilirubin < 1.25×ULN(Upper Limit Of Normal)
   * ALT < 2.5×ULN; ALT < 5×ULN ( If have liver metastases)
   * AST < 2.5×ULN; AST < 5×ULN ( If have liver metastases)
   * Serum creatinine < 1.25×ULN, and endogenous Cr clearance > 45 ml/min(Cockcroft-Gault Formula)
   * Cholesterol ≤ 1.5×ULN and triglyceride≤ 2.5×ULN
   * Left ventricular ejection fraction(LVEF): ≥ LLN(Lower Limit Of Normal) by Color Doppler Ultrasonography
8. Female: Child bearing potential, a negative urine or serum pregnancy test result 7 days before initiating famitinib.All subjects who are not surgically sterile or postmenopausal must agree and commit to the use of a reliable method of birth control for the duration of the study and for 8 weeks after the last dose of test article. Male: All subjects who are not surgically sterile or postmenopausal must agree and commit to the use of a reliable method of birth control for the duration of the study and for 8 weeks after the last dose of test article;
9. Patient has given written informed consent.

Exclusion Criteria:

1. More than one chemotherapy treatment regimen (except,either neoadjuvant or adjuvant or neoadjuvant plus adjuvant) for advanced and/or metastatic or recurrent NSCLC;
2. Previous therapy with other VEGFR inhibitors (including sunitinib,sorafenib,pazopanib,axitinib,other than bevacizumab) or docetaxel for treatment of NSCLC;
3. Radiographical evidence of cavitary or necrotic tumours;
4. Centrally located tumours with radiographical evidence (CT or MRI) of local invasion of major blood vessels;
5. Pre-existing ascites and/or clinically significant pleural effusion;
6. Pulmonary hemorrhage/ bleeding event ≥ CTCAE gr. 2 before initiating investigational drugs;
7. History of clinically significant haemoptysis within the past 3 months（24h >half teaspoon）;
8. Current peripheral neuropathy greater than CTCAE grade 2;
9. Other malignancy within the past 3 years other than basal cell skin cancer, or carcinoma in situ of the cervix;
10. Active brain metastases (such as stable time ≤ 4 weeks,no radiotherapy treatment,any symptoms,or seizures treatment needing) or leptomeningeal disease.;
11. Treatment with other investigational drugs or other anti-cancer therapy, or treatment in another clinical trial within the past 4 weeks before start of therapy or concomitantly with this trial;
12. Persistence of clinically relevant therapy related toxicities from previous chemotherapy and/or radiotherapy;
13. Treatment with cytotoxic drugs, radiotherapy(except extremities and brain) , immunotherapy , monoclonal antibody, or TKI inhibitor therapy within the past 4 weeks, being previous anti-cancer treatment interval ≤ 4 weeks.;
14. Patients with hypertension using combination therapy (systolic blood pressure>140 mmHg, diastolic blood pressure>90 mmHg). Patients with unstable angina, myocardial ischemia or myocardial infarction in the past 6 months, congestive heart failure>NYHA II,and arrhythmia (including QTcF interval ≥ 450ms for male and 470ms for female);
15. Urine protein ≥ + + and confirmed the 24-hour urinary protein>1.0 g;
16. History of major thrombotic or clinically relevant major bleeding event in the past 6 months，and known inherited predisposition to bleeding or thrombosis;
17. PT or APTT bias from normal range≥50%;
18. Application of anticoagulants or vitamin K antagonists such as warfarin, heparin or its analogues;If the prothrombin time international normalized ratio (INR) ≤ 1.5, with the purpose of prevention, the use of small doses of warfarin (1mg orally, once daily) ， low-dose aspirin (less than 100mg daily) is allowed;
19. Preexisting thyroid dysfunction, even using medical therapy, thyroid function cannot maintain in the normal range;
20. Diabetes mellitus can not controlled with hypoglycemic agent;
21. Active or chronic hepatitis C and/or B infection with liver dysfunction;
22. History of immunodeficiency disease, concurrent acquired or congenital immunodeficiency,or history of organ transplantation;
23. Serious infections requiring systemic antibiotic therapy;
24. Variety of factors that affect the oral medication (such as inability to swallow, gastrointestinal resection, chronic diarrhea and intestinal obstruction);
25. Significant weight loss (>10 %) within the past 6 months;
26. Pregnancy , breast feeding or child bearing potential, a positive urine or serum pregnancy test result 7 days before initiating famitinib;
27. Active alcohol or drug abuse;
28. Any contraindications for therapy with docetaxel；History of severe hypersensitivity reactions to docetaxel or other drugs formulated with polysorbate 80 (Tween 80)；Hypersensitivity to famitinib and/or the excipients of the trial drugs；Hypersensitivity to contrast media;
29. Psychological, familial, sociological, or geographical factors potentially hampering compliance with the study protocol and follow-up schedule;
30. Patients unable to comply with the protocol;
31. Evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of famitinib in combination with standard-dose docetaxel(60 mg/m^2) | 3 weeks
  MTD was defined as the highest dose at which incidence of dose-limiting toxicities(DLTs) in Cyle 1 was ≤33.3%(0/3,1/6,2/6)

SECONDARY OUTCOMES:
Incidences of Adverse Events according to Common Toxicity Criteria (CTC version 4.0) associated with increasing doses of famitinib | 1 years
Pharmacokinetics-AUC | 6 weeks
  Area under the plasma concentration-time curve (AUC) for famitinib and docetaxel
Pharmacokinetics-Cmax | 6 weeks
  Maximum measured plasma concentration (Cmax) for famitinib and docetaxel
Pharmacokinetics-Tmax | 6 weeks
  Time from dosing to the maximum plasma concentration (Tmax) for famitinib and docetaxel
Pharmacokinetics-t1/2 | 6 weeks
  Terminal half-life (t1/2(ss)) for famitinib and docetaxel
Objective Response Rate (ORR) | 6 weeks
Progress free survival (PFS) | 1 years

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China